CLINICAL TRIAL: NCT00424723
Title: A Phase II Study of Pemetrexed in Patients With Advanced Neuroendocrine Tumors
Brief Title: Pemetrexed in Patients With Advanced Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Responsible Party: Matthew Kulke, MD, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-309
Record Dates: First submitted 2007-01-18; First posted 2007-01-19 (Estimated); Last update posted 2010-08-12 (Estimated); Status verified 2010-08

CONDITIONS: Neuroendocrine Tumors
Keywords: pemetrexed; neuroendocrine tumors; metastatic neuroendocrine tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed — Given intravenously over 10 minutes every 21 days (21 days equals one cycle). Subjects will continue to receive pemetrexed as long as their disease does not worsen and they do not experience any serious side effects.

SUMMARY:
The purpose of this study is to find out what effects (good and bad) pemetrexed has on patients with advanced neuroendocrine tumors.

DETAILED DESCRIPTION:
* 1 cycle is equal to 21 days. Every 21 days the following will be performed: a review of the patients symptoms and medications; physical exam; blood tests; vital signs; and pemetrexed infusion.
* Every 3 cycles (9 weeks) an assessment of disease extent by CT scan and a 24 hour urine collection (if applicable) will be performed.
* Before patients start receiving pemetrexed, they will be given folic acid, vitamin B12 and dexamethasone to help reduce the chance of significant side effects. Dexamethasone will be taken the evening before, the morning before and the evening after receiving pemetrexed. Folic acid should be taken daily beginning 5-7 days before the first dose of pemetrexed and should be continued for three weeks after the last dose of pemetrexed. Vitamin B12 will be given as an injection 1-2 weeks before the first dose of pemetrexed and once every 9 weeks until 3 weeks after the last dose of pemetrexed.
* Patients can continue to receive treatment with pemetrexed unless there is evidence that their tumor has grown or they are experiencing serious side effects.
* Immediately after the patient has completed the study, they will be given a physical exam, including vital signs, a CT scan, and blood tets. The study staff will continue to monitor the patients health either by clinic visits or phone calls every three months for the remainder of your life.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or locally unresectable neuroendocrine tumor, excluding small cell carcinoma
* Measurable tumor
* 18 year of age or older
* ECOG performance status of 0,1 or 2
* Life expectancy of greater than 12 weeks
* WBC: > 3.0/mm3
* Plts: > 100,000/mm3
* Bilirubin: < 2.0 mg/dl
* AST < 3 x ULN (except in patients with known hepatic metastases wherein SST may be < 5 x ULN)
* Neutrophils > 1000/mm3
* Creatinine Clearance > 45 ml/min. Should be measured using the standard Cockroft-Gault formula

Exclusion Criteria:

* Prior treatment with pemetrexed
* Clinically apparent central nervous system metastases or carcinomatous meningitis
* Myocardial infarction in the past 6 months
* Major surgery in the past two weeks
* Uncontrolled serious medical or psychiatric illness
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2005-12; Primary Completion 2007-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To assess the radiologic response rate associated with pemetrexed in patients with neuroendocrine tumors. | 2 years

SECONDARY OUTCOMES:
To perform an analysis of the biochemical response rate | 2 years
to assess the toxicity associated with pemetrexed | 2 years
and to assess the progression-free and overall survival of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Kulke, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Center, Boston, Massachusetts, United States

REFERENCES:
- [Result] Chan JA, Zhu AX, Stuart K, Bhargava P, Earle CC, Clark JW, Casey C, Regan E, Kulke MH. Phase II study of pemetrexed in patients with advanced neuroendocrine tumors. Cancer Chemother Pharmacol. 2010 Oct;66(5):961-8. doi: 10.1007/s00280-010-1248-6. Epub 2010 Feb 4. PMID 20130879